CLINICAL TRIAL: NCT04888806
Title: Camrelizumab Combined With Microwave Ablation and Chemotherapy in the Treatment of Colorectal Cancer Liver Metastasis/Pulmonary Metastasis -a Single-arm Prospective Study
Brief Title: A Trial of Camrelizumab Combined With Microwave Ablation and Chemotherapy in the Treatment of Colorectal Cancer Liver Metastasis/Pulmonary Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yanqiao Zhang, Director, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-HLJ-019
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastases; Lung Metastases
MeSH Terms: interventions — camrelizumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+ablation +chemotherapy (Experimental): The enrolled patients received ablation of liver metastases/pulmonary metastasis first, followed by chemotherapy (standard treatment plan for advanced colorectal cancer, determined by the investigator) and camrelizumab treatment (200mg, iv, q3w) one week later. If the patient has multiple metastatic tumors, ablation therapy needs to be performed in multiple times. Sequential chemotherapy and camrelizumab is administered one week after each ablation therapy. Treatment will continue until disease progression, unacceptable toxicity, or voluntary patient withdrawal.
  Interventions: Drug: Camrelizumab; Procedure: ablation; Drug: chemotherapy

INTERVENTIONS:
Drug: Camrelizumab — d1，200mg, iv, q3w
Procedure: ablation — the 37 enrolled patients received ablation of liver/lung metastases ，If the patient has multiple metastatic tumors, ablation therapy needs to be performed in multiple times.
Drug: chemotherapy — standard treatment plan for mCRC, determined by the investigator

SUMMARY:
Currently, comprehensive treatments for liver metastasis/pulmonary metastasis that cannot reach NED include systemic chemotherapy, interventional chemotherapy, molecular targeted therapy, immunotherapy, and local treatments (ablation therapy, radiation therapy, etc.) for liver metastases. Combination therapy model of local ablation, systemic chemotherapy, and anti-PD -1 monoclonal antibody hopefully can prolong patient survival. This trial will evaluate the effectiveness and safety of carrelizumab combined with microwave ablation and chemotherapy in the treatment of colorectal cancer liver metastasis/pulmonary metastasis

DETAILED DESCRIPTION:
This is a phase II, single-arm prospective trial of local ablation combined with chemotherapy and camrelizumab for liver metastasis/pulmonary metastasis in colorectal cancer. The enrolled patients received ablation of liver metastases/pulmonary metastasis first, followed by chemotherapy (standard treatment plan for advanced colorectal cancer, determined by the investigator) and camrelizumab treatment (200mg, iv, q3w) one week later. If the patient has multiple metastatic tumors, ablation therapy needs to be performed in multiple times. Sequential chemotherapy and camrelizumab is administered one week after each ablation therapy. Treatment will continue until disease progression, unacceptable toxicity, or voluntary patient withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Two types of imaging or histology/cytology confirmed colorectal cancer patients with liver metastasis/lung metastasis ;
2. Must have CT or MRI examination for the past 3 months;
3. In addition to ablation lesions, there are measurable metastatic lesions (spiral CT scan ≥10mm, meet mRECIST 1.1 standard);
4. Expected survival time> 3 months;
5. Patients who have received at least one prior systemic treatment;
6. The damage caused by the subject receiving other treatments has been restored;
7. Known KRAS, NRAS, BRAF and HER2 gene status;
8. Age: 18 to 70 years old, no gender limit;
9. ECOG PS: 0-2 points;
10. The functions of vital organs meet the following requirements:

    1. .Absolute neutrophil count ≥1.5×109/L, platelet ≥100×109/L, hemoglobin

       ≥9g/dL;
    2. . Bilirubin ≤1.5 times ULN (can be included in patients drained by retrograde technique); ALT and AST

       ≤5 times ULN
    3. . Creatinine <120μmol/ L, or MDRD creatinine clearance rate> 60 mL/min
11. Women of childbearing age must have a negative pregnancy test (βHCG) before starting treatment, Women and men of childbearing age (have sex with women of childbearing age) must agree to use effective contraception during treatment and for 6 months after the last treatment dose is administered
12. Signature of patient information and informed consent

Exclusion Criteria:

1. Women who are pregnant or breastfeeding, or have fertility but refuse to take contraceptive measures;
2. Suffer from other malignant tumors within 5 years, except for fully treated cervical carcinoma in situ or skin squamous cell carcinoma, or skin basal cell carcinoma that has been basically controlled;
3. Those with uncontrolled, symptomatic brain metastases or a history of uncontrollable mental illness or severe intellectual or cognitive dysfunction;
4. Subjects with active, known or suspected autoimmune diseases, hypothyroidism requiring only hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss) Can be selected
5. Patients with active hepatitis B or C, chronic infection of hepatitis B virus (HBV) or hepatitis C virus (HCV) with a viral load of less than 500 IU/mL are allowed to participate in the study, but need to continue during the study period or start a full-course standardized antiviral treatment;
6. Congestive heart failure, uncontrollable arrhythmia, myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months; or other patients who cannot tolerate surgery;
7. Severe active infections that require intravenous antibiotic treatment occurred during the enrollment period;
8. Those who are allergic to test drugs;
9. Live vaccines have been vaccinated or will be vaccinated within 30 days before the administration of Camrelizumab;
10. Patients who cannot comply with the trial protocol or cannot cooperate with follow-up;
11. The researcher believes that it is inappropriate to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
12-month progression-free survival (PFS) | 1 year
  The date of first treatment until the date of progression using the RECIST 1.1 criteria, or death due to any cause,whichever comes first.

SECONDARY OUTCOMES:
Objective response rate(ORR) | 3 years
  ORR, which is defined as the proportion of subjects who achieve a best response of complete response(CR) or partial response (PR) using the RECIST 1.1 criteria.
Disease control rate (DCR) | 3 years
  DCR, which is defined as the proportion of subjects who achieve a response of complete response, partial response and stable disease (CR+PR+SD) in the total number of evaluable subjects using the RECIST 1.1 criteria.
progression-free survival (PFS) | 3 years
  The date of first treatment until the date of progression using the RECIST 1.1
Overall Survival(OS) | 3 years
  Overall Survival, defined from the date of first treatment to the date of death due to any cause.